CLINICAL TRIAL: NCT05445115
Title: DAT: Dyspareunia Alleviation Trial
Brief Title: The Mollie Study, a Study to Evaluate the Safety and Efficacy of the Mollie Medical Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: JSP Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP-01
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Dyspareunia
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Intervention Model Description: Treatment arm and sham arm
Who Masked: Participant
Masking Description: Subjects are blinded as to which arm they are participating in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Actual treatment device
  Interventions: Device: Mollie device
- Sham (Sham Comparator): Sham/placebo device
  Interventions: Device: Mollie device

INTERVENTIONS:
Device: Mollie device — medical device
  Other Names: Sham

SUMMARY:
Study to evaluate the use of a medical device in relieving collision dyspareunia

ELIGIBILITY:
Inclusion Criteria: Females 18 years of age and older with a diagnosis of collision dyspareunia -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Dyspareunia Alleviation | 12 weeks
  The Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v.4.0, Change from Baseline in Pain Scores on the Visual Analog Scale at 13 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vero Clinics, Decatur, Illinois, United States